CLINICAL TRIAL: NCT01000428
Title: The Role of PET During Erlotinib Treatment to See the Responsiveness of Tumor Early in Patients With Non-small Cell Lung Cancer
Brief Title: The Role of Positron Emission Tomography (PET) During Erlotinib Treatment for Non-small Cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Sang-We Kim/Professor, Asan Medical Center
Other Study IDs: AMC-2008-0511
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Last update posted 2009-10-27 (Estimated); Status verified 2009-10

CONDITIONS: Erlotinib; Lung Cancer
Keywords: NSCLC; Tarceva; Positron emission technology; FLT; FDG
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Erlotinib is an inhibitor of the epidermal growth factor receptor (EGFR) tyrosine kinase. Higher response rates were observed in a subset of patients with female gender, Asian ethnicity, no smoking history, mutations in EGFR tyrosine kinase, high EGFR gene copy number and adenocarcinoma histology. However, the therapeutic effect of Erlotinib is not confined to patients whose tumors harbor EGFR mutations and other predictors of efficacy of this agent. And these tests require time and sufficiently large specimens for processing, whereas many patients with advanced NSCLC are diagnosed based on cytology alone.

This study was designed to evaluate FLT-PET or FDG-PET usefulness in the early assessment of treatment response and in predicting patient outcome after erlotinib monotherapy for patients with non-small cell lung cancer prospectively. Changes in tumor FLT or FDG uptake 7 days after the initiation of treatment will be compared between responders and nonresponders based on subsequent CT scans.

DETAILED DESCRIPTION:
1. Primary objectives:

   To see whether the % change in SUVmax of a tumor with FLT-PET or FDG-PET at 7 days after initiating erlotinib treatment compared with baseline SUVmax (ΔSUVmax) would predict the tumor's responsiveness. And the responsiveness will be decided with the CT scan after 6 weeks of erlotinib treatment.
2. Secondary objectives:

To compare ΔSUVmax and the degree of tumor shrinkage in longest diameter during erlotinib treatment.

To see ΔSUVmax in the tumors with stable disease. To see the time to progression and overall survival according to ΔSUVmax. To compare the result of FDG-PET and FLT-PET.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* Histologically documented non-small cell lung cancer with metastasis (Stage IV) or locally advanced (Stage IIIB) with malignant effusion.
* At least 1 measurable lesion as defined by RECIST. All target lesions must have a unidirectional diameter of at least 1cm. Baseline measurements must be compared within 4 weeks prior to enrollment.
* ECOG PS 0-2
* At least 3 weeks since the 1st line systemic therapy regimen prior to enrollment. Patients must have recovered to NCI CTCAE v3.0 grade I from all toxicities. But 1st line erlotinib treatment is also allowed.
* At least 1 week since the last radiotherapy. Patients must have recovered from all acute toxicities from radiotherapy.
* Patients must have adequate hematologic, renal and liver function as defined by Hb > 9g/dL, neutrophils > 1000/mm3, platelets > 50,000/mm3, creatinine < 2mg/dL, and AST (SGOT) and/or ALT (SGPT) < 5 x UNL (upper normal limit).
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedures.
* Written and voluntary informed consent understood, signed and dated.

Exclusion Criteria:

* Prior EGFR TKI treatment.
* Symptomatic brain metastasis. Brain metastases stable < 2 weeks before dosing or requiring concurrent steroid treatment or with clinical symptoms.
* Major surgery within 3 weeks prior to study enrollment.
* Previous (less than 3 years ago) or current malignancies at sites other than curatively treated in situ carcinoma of cervix, or basal or squamous cell carcinoma of the skin.
* Severe medical illness or active infection that would impair the ability to receive erlotinib.
* Pregnancy or breast feeding.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically documented non-small cell lung cancer with metastasis (Stage IV) or locally advanced (Stage IIIB) with malignant effusion.
Sampling Method: Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-05 (Estimated); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, SongPa-Gu, South Korea